CLINICAL TRIAL: NCT03930693
Title: Investigation of the Oral Microbiome in Pregnancy - do Differences in Oral Bacterial Profiles and Nitrate Metabolism Contribute to Blood Pressure Regulation in Pregnant Women?
Brief Title: Role of the Oral Microbiome in Blood Pressure Regulation in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Dr Jenny Myers, Principal Investigator, University of Manchester
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 246813
Record Dates: First submitted 2019-04-23; First posted 2019-04-29 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Gestational Hypertension
Keywords: Pregnancy; hypertension; nitrate; beetroot juice
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension

STUDY DESIGN:
Intervention Model Description: Beetroot juice intervention given to all participants (1 dose only)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normotensive pregnant women (Experimental): Normotensive pregnant women
  Interventions: Dietary Supplement: Beetroot juice
- Hypertensive pregnant women (Experimental): Hypertensive pregnant women
  Interventions: Dietary Supplement: Beetroot juice
- Normotensive non-pregnant women (Experimental): Normotensive non-pregnant women
  Interventions: Dietary Supplement: Beetroot juice
- Hypertensive non-pregnant women (Experimental): Hypertensive non-pregnant women
  Interventions: Dietary Supplement: Beetroot juice

INTERVENTIONS:
Dietary Supplement: Beetroot juice — Beetroot juice shot (70mL containing 400mg inorganic nitrate)

SUMMARY:
High blood pressure in pregnancy is associated with poor outcomes for both mum and baby, increasing the risk of pregnancy complications including pre-eclampsia, fetal growth restriction and preterm birth. The development of new blood pressure lowering interventions suitable for use in pregnancy is a key research priority.

Inorganic nitrate is a compound found in certain types of food, particularly green leafy vegetables and beetroot. Nitrate provides an important source of nitric oxide (NO), a molecule involved in keeping blood vessels healthy and regulating blood pressure. Supplementation with nitrate in the diet, using interventions such as beetroot juice, has been shown to reduce blood pressure and improve blood vessel function.

In order for dietary nitrate to have these beneficial effects, it needs to be converted in the body to nitrite, via bacteria that live in the mouth (oral bacteria). Differences in oral bacteria, and how they metabolise nitrate, are thought to influence blood pressure regulation and potentially response to dietary nitrate supplementation.

This study aims to understand (1) whether pregnant women with high blood pressure have a different composition of oral bacteria compared to healthy pregnant women and women who are not pregnant, and (2) how differences in oral bacteria affect blood pressure responses to a dose of dietary nitrate (in the form of beetroot juice).

ELIGIBILITY:
Inclusion Criteria:

* Normotensive or hypertensive women (hypertension as systolic blood pressure >140 mmHg and/or diastolic blood pressure >90 mmHg OR on anti-hypertensive medication)
* For pregnant women, between 20-28 weeks gestation

Exclusion Criteria:

* Multi-fetal pregnancy (for pregnant women)
* Age under 16, or over 45 years of age
* Lacking ability to consent
* Pre-existing diabetes (Type 1/Type 2)
* Previous history of pre-term FGR (delivery before 32 weeks with FGR)
* Current tobacco smoker
* Body Mass Index greater than or equal to 40 or less than or equal to 18
* Use of any of the following drugs in the last 6 months: systemic antibiotics, antifungals, antivirals or antiparasitics (intravenous, intramuscular, or oral)
* Large doses of commercial probiotics (greater than or equal to 108 cfu or organisms per day) including tablets, capsules, lozenges, chewing gum or powders (ordinary dietary components such as yoghurts do not apply)
* Evidence of oral disease, assessed on screening proforma (current conditions of: oral candidiasis (thrush); Dental caries (tooth decay); Halitosis; Oral ulcerations/mouth ulcers; Wisdom tooth pain; Chronic dry mouth)
* Allergy to beetroot juice or lemon juice (both contained within the juice shot)

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Quantity of oral nitrate reducing bacterial species | Baseline
  Assessment of oral bacterial profile using next-generation sequencing (bacterial 16S rRNA sequencing)
Oral bacterial nitrate reductase activity | Baseline
  Assessment of oral nitrate reductase activity, measured using enzyme assay
Difference between groups in nitrate/nitrite concentrations before and after dietary nitrate dose | Baseline to 2.5 hour post-nitrate dose
  Measurement of plasma and salivary nitrate and nitrite concentrations, using high-performance liquid chromatography (HPLC)

SECONDARY OUTCOMES:
Difference between groups in blood pressure response to dietary nitrate dose | Baseline to 2.5 hour post-nitrate dose
  Change in blood pressure

OTHER OUTCOMES:
Correlation between salivary nitrate reductase activities and the change in salivary/plasma nitrite concentrations post-nitrate dose | Baseline to 2.5 hour post-nitrate dose
  Change in nitrite vs. baseline nitrate reductase activity
Correlation between changes in plasma nitrite concentrations and blood pressure lowering post-nitrate dose | Baseline to 2.5 hour post-nitrate dose
  Change in plasma nitrite vs. change in blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Myers, BM, PhD, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Maternal and Fetal Health Research Centre, St Mary's Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Willmott T, Ormesher L, McBain AJ, Humphreys GJ, Myers JE, Singh G, Lundberg JO, Weitzberg E, Nihlen C, Cottrell EC. Altered Oral Nitrate Reduction and Bacterial Profiles in Hypertensive Women Predict Blood Pressure Lowering Following Acute Dietary Nitrate Supplementation. Hypertension. 2023 Nov;80(11):2397-2406. doi: 10.1161/HYPERTENSIONAHA.123.21263. Epub 2023 Sep 13. PMID 37702047